CLINICAL TRIAL: NCT06502002
Title: Dexmedetomidine Infusion and Postoperative Lung Aeration After Thoracic Surgery: A Randomized, Placebo-Controlled Pilot Trial
Brief Title: Dexmedetomidine Infusion and Postoperative Lung Aeration After Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Matthew B. Allen, MD, Staff Anesthesiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023P001017
Record Dates: First submitted 2023-08-31; First posted 2024-07-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Surgery-Complications; Respiratory Complication; Lung Injury, Acute
Keywords: dexmedetomidine; lung ultrasound; lung resection; thoracic surgery; aeration
MeSH Terms: conditions — Acute Lung Injury | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This will be a randomized, placebo-controlled, double-blinded, pilot trial with two parallel groups (1:1 ratio) receiving either dexmedetomidine) or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Dexmedetomidine or placebo infusion will be blinded (by pharmacist preparing the study drug) to the patient, treating physicians, and investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine infusion arm
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Placebo (Placebo Comparator): Normal saline infusion arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Initial dexmedetomidine bolus of 1 mcg/kg over 30 min after induction, followed by an infusion rate of 0.3 mcg/kg/hr that will be stopped 30-45 minutes before the end of the surgery or once a maximum dose of 2mcg/kg has been achieved, whichever comes first.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Placebo — normal saline infusion
  Arms: Placebo

SUMMARY:
This will be a randomized, placebo-controlled, double-blinded, pilot trial with two parallel groups (1:1 ratio) receiving either dexmedetomidine (initial bolus of 1 mcg/kg over 30 min after induction, followed by an infusion rate of 0.3 mcg/kg/hr that will be stopped 30-45 minutes before the end of the surgery or upon reaching maximum dose of 2mcg/kg, whichever comes first) or placebo (normal saline as a bolus followed by maintenance infusion at the same rate of the intervention group).

Dexmedetomidine is frequently administered in thoracic surgery. Using local data from the Brigham and Women's Hospital, dexmedetomidine was used in a third of the thoracic procedures performed over the past three years. However, there is no consensus as to the optimal protocol of administration, therefore clinical practice is highly heterogeneous (bolus versus continuous infusion) and mostly depends on the preferences of anesthesia providers. In our institution, the dose of dexmedetomidine is typically 0.5 mcg/kg but varies based on attending preferences and experience. Given the heterogenous practices in dexmedetomidine administration, one of the objectives is to assess the feasibility of adhering to a dexmedetomidine protocol using an initial loading dose of 1 mcg/kg over 30 minutes after induction followed by a continuous infusion of 0.3 mcg/kg/hr. The infusion will stop 30-45 minutes prior to the end of surgery or once a maximum dose of 2mcg/kg has been achieved, whichever comes first. The control group will receive normal saline (similar bolus followed by maintenance infusion at the same rate of the intervention group).

DETAILED DESCRIPTION:
Dexmedetomidine is an opioid-sparing anesthetic with minimal effect on adaptive physiologic processes such as respiratory drive and hypoxic pulmonary vasoconstriction (HPV). Recent translational research has demonstrated that dexmedetomidine is associated with less alveolar inflammation and better respiratory mechanics in thoracic surgery under one-lung ventilation (OLV). However, it is unclear whether such results translate into better postoperative lung aeration and superior pulmonary outcomes. Several biological mechanisms have been postulated to explain the lung protective effects of dexmedetomidine. Based on experimental models under OLV, dexmedetomidine has been shown to minimize mechanical ventilation-induced lung injury through the inhibition of inflammatory pathways, thus enhancing pulmonary function recovery, improving respiratory mechanics, and potentially preventing postoperative pulmonary complications (PPCs). There is also clinical evidence to suggest dexmedetomidine may improve respiratory mechanics as well as prevents non-cardiopulmonary complications such as acute kidney injury (AKI) in adult cardiac surgical patients, as well as delirium in both cardiac and non-cardiac patients.

The research group from the BWH anesthesia department recently conducted a meta-analysis about the current evidence on dexmedetomidine in thoracic surgery, demonstrating beneficial effects in atelectasis and hypoxemia with low to moderate certainty. Unfortunately, current trials on this topic have limited sample size, and do not provide accurate and standardized outcome measurements. Dexmedetomidine has been shown to have organ protection properties, but there is no conclusive evidence to support its use for pulmonary protection in thoracic surgery. This trial would be the first to demonstrate an effect of dexmedetomidine on the trajectory of postoperative lung aeration and diaphragmatic excursion measured by ultrasound. Furthermore, the feasibility of a large, randomized controlled trial on dexmedetomidine for the prevention of pulmonary complications in thoracic surgery will be assessed. It is important to note that all the trials conducted on this topic have been conducted in Asia (limiting its generalizability), are relatively small (sample size of 30-50 patients) and have studied mainly respiratory mechanics.

Postoperative pulmonary complications are relatively common among patients undergoing thoracic surgery. The development of PPCs raises hospital costs (5,000-10,000 USD), prolong length of hospital stay (2-3 days), and affects quality of recovery. Similarly, lung aeration loss is considered a subclinical characteristic of lung injury induced by OLV, which can persist for several days after thoracic surgery. Several protective ventilatory strategies have been proposed to prevent PPCs, such as low tidal volume (TV) (i.e., TV [< 6mL/kg] and alveolar recruitment), yet the literature shows conflicting results, and the incidence of pulmonary complications continues to occur. Therefore, it is imperative to study and implement novel, pharmacologic lung protective interventions in thoracic surgery for the prevention of lung aeration loss and subsequent pulmonary complications.

In this study protocol, dexmedetomidine is postulated as an adjunct with possible pulmonary clinical benefits. Previous evidence suggests a possible effect on atelectasis, hypoxemia, and pneumonia, but the certainty of the evidence is low to moderate. Undertaking a pilot trial on dexmedetomidine and lung aeration in thoracic surgery would be useful to assess the feasibility for a large, randomized trial.

2. Specific Aims and Objectives

Objective #1: To determine the feasibility of a trial assessing the effect of dexmedetomidine administration on postoperative lung aeration after thoracic surgery.

Objective #2: To compare the effect of dexmedetomidine administration protocol versus placebo on postoperative lung aeration and diaphragmatic excursion measured by lung ultrasound.

Objective #3: To evaluate the adherence to a protocol of dexmedetomidine administration during thoracic surgery under one-lung ventilation.

3. General Description of Study Design

This will be a randomized, placebo-controlled, double-blinded, pilot trial with two parallel groups (1:1 ratio) receiving either dexmedetomidine (initial bolus of 1 mcg/kg over 30 min after induction, followed by an infusion rate of 0.3 mcg/kg/hr that will be stopped 30-45 minutes before the end of the surgery or once a maximum dose of 2mcg/kg has been achieved, whichever comes first) or placebo (normal saline as a bolus followed by maintenance infusion at the same rate of the intervention group).

Dexmedetomidine is frequently administered in thoracic surgery. Using local data from the Brigham and Women's Hospital, dexmedetomidine was used in a third of the thoracic procedures performed over the past three years. However, there is no consensus as to the optimal protocol of administration, therefore clinical practice is highly heterogeneous (bolus versus continuous infusion) and mostly depends on the preferences of anesthesia providers. At the Brigham and Women's Hospital, the dose of dexmedetomidine is typically 0.5 mcg/kg but varies based on attending preferences and experience. Given the heterogenous practices in dexmedetomidine administration, one of the objectives is to assess the feasibility of adhering to a dexmedetomidine protocol using an initial loading dose of 1 mcg/kg over 30 minutes after induction followed by a continuous infusion of 0.3 mcg/kg/hr. The infusion will be stopped 30-45 minutes prior to the end of surgery or once a maximum dose of 2mcg/kg has been achieved, whichever comes first. The control group will receive normal saline (similar bolus followed by maintenance infusion at the same rate of the intervention group).

4. Subject Selection

Inclusion criteria:

• Adult patients (Age >18 years until 80 years) undergoing lobectomy and/or segmentectomy.

Exclusion Criteria:

* Urgent or emergency thoracic surgery.
* Other concomitant non-pulmonary procedures (pleurectomy, diaphragmatic procedures, pericardiocentesis, esophageal procedures, thymectomy).
* Prior lung resection surgery.
* Epidural block for intraoperative or postoperative analgesia.
* Preoperative arrhythmia (first or second degree AV block without pacemaker) or significant bradycardia (heart rate < 50).
* Preoperative hypotension (mean arterial blood pressure < 65 mmHg).
* Severe functional liver or kidney disease.
* Non-English speakers
* Consent withdrawal.

Identification of individuals will be completed every day through Epic. The list of thoracic surgeries will be reviewed each day by one of the co-investigators. Individuals will be contacted via phone 24-48 hours prior to the surgery for pre-screening questions and to determine their interest in participating in the study. Individuals will be consented on the day of surgery at the preoperative area by one of the co-investigators.

Women and minorities will be represented in this study and will reflect the thoracic surgery population at Brigham and Women's Hospital (BWH) undergoing the eligible procedures. Based on prior studies conducted on this patient population, we estimate that the sample population will be 57% women, approximately 6% African American, 5% Asian, and 11% Latino. Patients over 65 years old comprise 52%, and low-income population is 4%. The investigators will make every effort to ensure proportional representation by sex/gender, race, and ethnicity (subjects are a sample of thoracic surgical patients), so the investigators do not expect significant deviations from these estimates.

5. Subject Enrollment

Allocation of individuals to the groups will be performed using a predetermined randomized sequence, which will be generated using the asymptotic maximal procedure (https://ctrandomization.cancer.gov/about/). Eligible patients will be contacted via phone call within 24-48 hours prior to surgery for pre-screening questions and assess possible participation in the study. On the day of surgery, the participant will be approached by one of the investigators who will explain further details of the trial and provide an electronic informed consent (e-Consent) on a tablet.

6. STUDY PROCEDURES

Pharmacy will be contacted the day before to start processing the study drug based on the randomization list. A research collaborator will collect intraoperative information prospectively, including time to start study drug, time of lung isolation, time of two lung ventilation, respiratory mechanics, and compliance with administration protocol. In the postoperative period, patients will be followed up for 2 days. In the PACU, an investigator will scan anterior, lateral, and posterior quadrants of both lungs, estimate the lung ultrasound score (see Appendix), and save the images. A second independent investigator will estimate the scores independently. Serial assessments will be performed preoperatively (in the preoperative area), immediately after surgery in the recovery area, and at postoperative days 1 and 2. The assessment of complications will end at post-operative day 30. Safety outcomes and pulmonary complications will be collected by another blinded investigator.

Primary outcome:

• Lung aeration score measured by ultrasound at the post-anesthesia care unit (PACU) as described by Monastesse et al. Serial assessments will be performed at postoperative days 1 and 2 (POD1 and POD2): time frame of measurements 2 days.

Secondary outcomes:

* Diaphragmatic dysfunction: defined as a diaphragmatic excursion < 1cm
* Intraoperative hypoxemia (SpO2 < 90%)
* Postoperative atelectasis (radiographic evidence of lung collapse: descriptive parameter)
* Pneumonia

  - radiologic evidence of consolidation (descriptive parameter),

  - fever (temperature T>38.5C)
  * white cell count (WBC) > 10G/L.
* Acute respiratory distress syndrome (ARDS) - PaO2/FiO2 <200

  - acute onset
  * bilateral lung infiltrates on chest radiograph
  * absence of heart failure
* Pulmonary edema (clinical description from chest radiograph
* Reintubation. - Timeframe for assessment of complications: 30 days.

  7. Risks and Discomforts

Protection Of Human Subjects

- Human Subject Involvement and Characteristics There is a risk of breach of confidentiality with individually identifiable health information. The database will have de-identified data using an assigned ID on all study related documents. Once the patient consents to the protocol, he or she will be assigned a unique patient identifier number. As a result, the study database will hold strictly de-identified data using an arbitrary participant ID; paper forms will be stored in a secure location and referenced only for scheduling contacts; and a bridging table associating the two entities will be stored in yet another secure location.

Upon initiating the study, all data will be collected and processed using rigorous quality-control methods. As the data forms are completed, they will be entered by the research staff into the secure access de-identified database. All paper forms will be stored in a locked cabinet in a locked room in a secure building. Neither the name of the patient nor any other personally identifying information will be used in any reports or publications that result from this study.

Potential Risks:

The study will not alter the surgeon's or patient's plan for surgery. A participant may be at risk if they have an adverse reaction to the medication (dexmedetomidine). Dexmedetomidine has been reported to have the following clinical side effects:

* Bradycardia
* Hypotension
* Somnolence

  8. Benefits Increasing understanding of the possible lung protective mechanisms of dexmedetomidine.

Patients in the dexmedetomidine group may also benefit from better pain control given the long-acting analgesic effects of dexmedetomidine.

9. Statistical Analysis

An exploratory analysis of baseline demographic and clinical characteristics will be performed. Compliance with the protocol of dexmedetomidine and/or placebo will be calculated as a percentage of complete adherence to the administration of either solution as stated above. Feasibility will be defined as a compliance greater than 80%. Both groups will be compared in terms of lung ultrasound score in each side (operative vs non-operative) of the thorax at PACU, and postoperative days 1 and 2. Similarly, secondary outcomes (diaphragmatic dysfunction, pulmonary complications) will be compared between both groups. Our analysis will be adjusted for multiple testing hypothesis. The estimated sample size is 100 patients (50 patients in each group) assuming a mean LUS of 14 vs 11 between the control and intervention groups, respectively, with a standard deviation of 5, a missing follow-up of 10%, an alpha error of 0.05, and 80% power. All statistical analyses will be performed in Stata v14.0 (College Station, TX, USA).

Analysis:

Continuous variables will be reported as means ± standard deviation (SD) or median with their corresponding interquartile ranges based on the distribution of the data, which will be determine using Kolmogorov test. Dichotomous variables will be reported as numbers (percentages). Between-group comparisons of continuous variables will be performed using the independent Student t test. P values < 0.05 will be considered statistically significant. Descriptive statistics will be used to report patient demographics and baseline characteristics.

Proportion of participants with postoperative pulmonary complications during admission will be reported (units: percentage). This will be extracted from the patient's electronic medical health records by a co-investigator.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients (Age >18 years until 80 years) undergoing lobectomy and/or segmentectomy.

Exclusion Criteria:

* Urgent or emergency thoracic surgery.
* Other concomitant non-pulmonary procedures (pleurectomy, diaphragmatic procedures, pericardiocentesis, esophageal procedures, thymectomy).
* Prior lung resection surgery.
* Epidural block for intraoperative or postoperative analgesia.
* Preoperative arrhythmia (second degree AV block or pacemaker) or significant bradycardia (heart rate < 50).
* Preoperative hypotension (mean arterial blood pressure < 65 mmHg).
* Severe functional liver or kidney disease.
* Non-English speakers
* Consent withdrawal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Lung aeration | 2 days
  Lung aeration score measured by ultrasound at the post-anesthesia care unit (PACU) as described by Monastesse et al. Serial assessments will be performed at postoperative days 1 and 2.

SECONDARY OUTCOMES:
Diaphragmatic dysfunction: defined as a diaphragmatic excursion < 1cm | 2 days
  diaphragmatic excursion measured by ultrasound
Intraoperative hypoxemia (SpO2 < 90%) | 1 day
  intraoperative hypoxemia measured by pulse oximetry
Postoperative atelectasis | 30 days
  radiographic evidence of lung collapse
Pneumonia | 30 days
  diagnosed by chest radiography (consolidations/opacifications), clinical or laboratory signs of infection
Acute Respiratory Distress Syndrome (ARDS) | 30 days
  Berlin Criteria (hypoxemia, sudden onset, absence of heart failure, bilateral infiltrates on chest radiograph)
Pulmonary edema | 30 days
  from chest radiograph (cephalization of vessel, diffuse opacification)
Reintubation | 30 days
  intubation of the trachea, application of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Allen, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dell'Aquila P, Raimondo P, Racanelli V, De Luca P, De Matteis S, Pistone A, Melodia R, Crudele L, Lomazzo D, Solimando AG, Moschetta A, Vacca A, Grasso S, Procacci V, Orso D, Vetrugno L. Integrated lung ultrasound score for early clinical decision-making in patients with COVID-19: results and implications. Ultrasound J. 2022 Jun 1;14(1):21. doi: 10.1186/s13089-022-00264-8. PMID 35648278